CLINICAL TRIAL: NCT02637284
Title: Phase I, Pilot Study in Healthy Volunteers, to Assess the Safety and Pharmacokinetics of PCO-02, Which Active Ingredient is BPC-157, a Penta-deca-peptide From Gastric Source.
Brief Title: PCO-02 - Safety and Pharmacokinetics Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PharmaCotherapia d.o.o. (Industry)
Collaborators: Hospital Ángeles Tijuana (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPK-1A/B-1.3
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — BPC 157

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Intervention 1a (cohort 1) (Experimental): Single dose of 1 oral tablet of PCO-02 containing 1 mg of Bepecin (12 subjects)
  Interventions: Drug: Bepecin
- Intervention 1a (cohort 2) (Experimental): Single dose of 3 oral tablets of PCO-02 containing 1 mg of Bepecin (12 subjects)
  Interventions: Drug: Bepecin
- Intervention 1a (cohort 3) (Experimental): Single dose of 6 oral tablets of PCO-02 containing 1 mg of Bepecin (12 subjects)
  Interventions: Drug: Bepecin
- Control group 1a (cohort 1) (Placebo Comparator): Single dose of 1 oral tablet of PCO-03 as placebo (2 subjects)
  Interventions: Drug: Placebo
- Control group 1a (cohort 2) (Placebo Comparator): Single dose of 3 oral tablets of PCO-03 as placebo (2 subjects)
  Interventions: Drug: Placebo
- Control group 1 a (cohort 3) (Placebo Comparator): Single dose of 6 oral tablets of PCO-03 as placebo by mouth (2 subjects)
  Interventions: Drug: Placebo
- Intervention 1b (Experimental): Multiple dose regime of 3 oral tablets of PCO-02 containing 1 mg Bepecin every 8 hours during 2 weeks (36 subjects)
  Interventions: Drug: Bepecin
- Control group 1b (Placebo Comparator): Multiple dose regime of 3 oral tablets of PCO-03 as placebo every 8 hours during 2 weeks (6 subjects)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bepecin — Phase 1a: Healthy volunteers will take a single dose of 1, 3 or 6 tablets by mouth of PCO-02 containing 1 mg of Bepecin to study safety and pharmacokinetics.
  Phase 1b: All subjects will take 3 tablets of PCO-02 containing 1 mg of Bepecin every 8 hours during two weeks, to study safety and pharmacokinetics.
  Other Names: PCO-02, BPC-157
  Arms: Intervention 1a (cohort 1); Intervention 1a (cohort 2); Intervention 1a (cohort 3); Intervention 1b
Drug: Placebo — Phase 1 a: Healthy volunteers will take a single dose of 1, 3 or 6 tablets by mouth of PCO-03 (placebo) as a control group.
  Phase 1b: All subjects will take 3 tablets of PCO-03 (placebo) every 8 hours during two weeks, as a control group.
  Other Names: PCO-03
  Arms: Control group 1 a (cohort 3); Control group 1a (cohort 1); Control group 1a (cohort 2); Control group 1b

SUMMARY:
Phase I clinical trial in healthy volunteers to study safety and pharmacokinetics of BPC-157, a pentadecapeptide from gastric source.

DETAILED DESCRIPTION:
Title: Phase I, pilot study in healthy volunteers, to assess the safety and pharmacokinetics of PCO-02, which active ingredient is BPC-157, a pentadecapeptide from gastric source.

Protocol Number: BPC-1A/B-1.2

Phase: I

Population: Healthy subjects, males or females, between 18 and 35 years of age.

Number of Sites: Single center, to be performed at Hospital Angeles, Tijuana.

Duration of Study: Six months, from January 01, 2015 to Jun 30, 2015.

Duration of Subject Participation: Three weeks

Intervention description:The study consists of the oral administration of PCO-02 tablets, each containing 1mg of BPC-157 or placebo. There will be two different administration schemes, which have been labeled as Phase 1a and Phase 1b.

* Phase 1a: Single dose administration of 1, 3 or 6 tablets of PCO-02 or placebo.
* Phase 1b: Oral administration of 3 tablets of PCO-02 or placebo three times daily for 2 weeks.

Study Goals:General: To assess, in healthy volunteers, the safety and pharmacokinetics of the oral administration of PCO-02, which pharmacological active product is BPC-157.

* Primary: To assess the safety of the oral administration of BPC-157.
* Secondary: To document the pharmacokinetics of BPC-157 after oral administration.

Study Design: This is a phase-I, randomized, placebo controlled, pilot study, in which a group of 42 healthy volunteers will receive orally an active compound (PCO-02) or placebo (PCO-03) to assess safety and pharmacokinetics.

Phase 1a: There will be three cohort groups, with 14 subjects each, that will receive a single oral dose of 1, 3 or 6 tablets of PCO-02, respectively or a similar dose of placebo (PCO-03). Randomization will be at a PCO-02-to-placebo ratio of 6:1 on each group, keeping a balance between men and women among groups.

For this phase, subjects will be admitted to the hospital for 24 hours and will be kept fasting before and after the administration of the study medication. Serial blood and urine samples will be obtained to document pharmacokinetics of BPC-157 peptide and the subjects from all groups will be observed for AE in order to determine the study medication's safety. A week after, subjects will return for clinical assessment and laboratory blood work to continue monitoring for AE's.

Also, the cohort that will receive 3 tablets will receive a second dose in a similar manner but after having had a meal.

Phase 1b:This second phase will initiate only once all subjects from prior phase have completed at least one week of follow-up and that there have been no SAE's related to study medication from phase 1a.

All of subjects from phase 1a will receive a single dose of 3 tablets of PCO-02 or placebo three times daily for a period of 14 days. The assignment to active (PCO-02) or placebo (PCO-02) will be the same as per the randomization for phase 1a.

This phase will be performed on an ambulatory manner, with the subjects being required to return to the clinic at days 0, 7 and 14 for safety and pharmacokinetics assessment.

Estimated Time to Complete Enrollment: One month

Study Goals:

Primary: Safety of oral administration of PCO-02, evaluated thru the systematic monitoring for adverse events during follow-up.

Secondary: Pharmacokinetics of oral BCP-157 (Tmax, Cmax, T1/2, AUC)

Clinical Assessment During Follow- Up: During phase 1a, subjects will be admitted to the hospital for 24 hours for monitoring adverse events and serial blood and urine sampling after a single dose of PCO-02 or placebo (PCO-03). Subjects will be discharged from the hospital on the next morning and will return a week after the initial dose for clinical assessment and laboratory blood work to continue monitoring for possible AE's. The first cohort will receive 1 tablet of PCO-02 or placebo. Increasing to the next dose requires the absence of severe adverse events related to the intervention in the previous dose cohort at one week of follow-up.

If there has been no AE's related to study medication, phase 1b will be started. Initial assessment of phase 1b will be the same as the final evaluation of phase 1a. All the subjects from phase 1a will receive a single dose of 3 tablets of PCO-02 three times daily, or a similar dose of placebo (PCO-03), for a period of 2 weeks. The assignment to active compound or placebo will be the same as for phase 1a.

The subject will be required to return to the clinic at days 7 and 14 for clinical, pharmacokinetics and safety assessment, including blood and urine sampling.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, between the ages of 18 and 35 years old.
* Willing and able to provide informed consent.
* Body Mass Index between 18.5 and 24.9 (normal)
* Normal blood work, according to following criteria: Leucocytes >3,000; Platelets >100,000; Hemoglobin >10.0 g/dL; AST, ALT and bilirubin < 2 times UNL; Creatinine < 2 times UNL.
* Normal ECG and chest x-rays, at the discretion of the cardiologist and radiologist, respectively.
* Negative urine pregnancy test (Women in childbearing age, sexually active).
* Willing to return for follow-up as required by the study.

Exclusion Criteria:

* History of psychiatric condition.
* Pregnant or lactating women.
* Clinically significant abnormalities on the ECG.
* Presence of medical or social conditions that, in opinion of the investigator, may prevent the proper participation of the volunteer subject in the study or in the assessment of its outcomes.
* Presence of an active systemic infection.
* Subjects receiving medical treatment for any medical condition, either acute or chronic.
* Recent (< 6 months) major surgery.
* Recent (< 1 year) alcohol abuse or illegal drug use.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Six months
  Any adverse event reported during the study.

SECONDARY OUTCOMES:
Maximum plasma concentration | 168 hours
  Cmax
Time to maximum plasma concentration | 168 hours
  Tmax
Area under the curve | 168 hours
  AUC
Elimination half life | 168 hours
  T1/2

CONTACTS AND LOCATIONS:
Overall Officials: Rufino Menchaca, PhD, Principal Investigator — Hospital Ángeles Tijuana
Locations (1):
- Hospital Ángeles Tijuana, Tijuana, Estado de Baja California, Mexico

REFERENCES:
- See also: Bepecin general information — http://www.ncbi.nlm.nih.gov/pubmed/?term=bpc+157